CLINICAL TRIAL: NCT05052762
Title: Comparison of the Effect of Weighted and Elastic Resistance Training of Gluteus Maximus in Subjects With Sacroiliac Joint Dysfunction
Brief Title: Effects of Weighted and Elastic Resistance Training of Gluteus Maximus in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01070 Aiman Mazhar
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Sacroiliac Disorder
Keywords: gluteus maximus; Elastic resistance training; weighted resistance training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Elastic resisted training for Gluteus Maximus strength. (Experimental): bilateral bridge, unilateral bridge, and non-weight-bearing hip extension in prone with the knee flexed at 90 degrees. In the next five sessions, abduction and external rotation in a quadruped and weight-bearing hip extension are added.
  Interventions: Other: Group A: Elastic resisted training for Gluteus Maximus strength
- Group B: Weight resisted training for Gluteus Maximus strength (Experimental): Prone hip extension with knee flexion against weighted resistance
  Interventions: Other: Group B: Weight resisted training for Gluteus Maximus strength

INTERVENTIONS:
Other: Group A: Elastic resisted training for Gluteus Maximus strength — Subjects attended physical therapy two times per week for a total of 10 visits. In the first five sessions, subjects performed the following exercises to strengthen the gluteus maximus: bilateral bridge, unilateral bridge, and non-weight-bearing hip extension in prone with the knee flexed at 90 degrees. In the next five sessions, abduction and external rotation in a quadruped ("fire hydrant" exercise) and weight-bearing hip extension (known as "deadlift" exercise) are added. Each exercise was performed for 10 repetitions. Elastic resistance was Added to the fire hydrant, hip extension in prone and deadlift exercises to allow each subject to perform at a 10-repetition maximum. The resistance for each subject was adjusted weekly as needed. The exercise program was performed under direct supervision only during the physical therapy sessions.
  Arms: Group A: Elastic resisted training for Gluteus Maximus strength.
Other: Group B: Weight resisted training for Gluteus Maximus strength — Subjects attended p two times per week for a total of 10 visits. The participants performed PHEKF in 90° knee flexion with 30° hip abduction and 10° hip extension to increase the muscle activity of the gluteus maximus. In the prone position, the participant performed 10° hip extension until the posterior knee reached the horizontal bar. The participants maintained 90° knee flexion with 30° hip abduction and 10° hip extension in the prone position against the resistance. Sandbags (3 kg) will be used to provide resistance on the ankle through a rope and pulley. Each subject performed three sets with three repetitions of five seconds each. 1-minute break is allowed between each set.
  Arms: Group B: Weight resisted training for Gluteus Maximus strength

SUMMARY:
This research aims to compare the effect of weighted and elastic resistance training of gluteus maximus in subjects with sacroiliac joint dysfunction. Randomized clinical trials were done. The sample size was 54. The subjects were divided into two groups, 27 subjects in the weighted resistance training group and 27 in the elastic resisted training group. The study duration was of 1 year. The sampling technique applied was the non-probability connivance sampling technique. Only 20-40 years of symptomatic subjects with pain in the SI region for at least 12 weeks (chronic) and had no previous physical therapy treatment were included. Tools used in the study are numeric pain scale, dynamometer, and Oswestry disability index. Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction or sacroiliitis are common terms used to describe the pain of the sacroiliac joint. It is usually caused by abnormal motion (i.e. hyper- or hypo-mobile) or mal-alignment of the sacroiliac joint. Sacroiliac joint (SI) dysfunction is a well-documented clinical entity that can cause pain and loss of function, The sacroiliac joint (SIJ) has been implicated as the primary pain source in 10% to 25% of the patients with low back pain. During pregnancy, 20% to 80% of the women experience low back or posterior pelvic pain frequently arising from the SIJ.

The Gluteus maximus is inserted proximally into the sacrum, the dorsal sacral ligaments, the posterior portion of the crest of the ilium, and the sacrotuberous ligament. The muscle fibers run inferiorly and laterally to the distal insertion, where it splits into two components. The upper half of the muscle inserts into the iliotibial tract of the fascia and the lower half into the gluteal tuberosity of the femur. Due to its attachments, the gluteus maximus is primarily involved in hip extension and lateral rotation.

Fischer & Houtz found in electromyography (EMG) study that the strongest contractions of gluteus maximus occurred with muscle setting by isometric contraction, external rotation, abduction with resistance, and vigorous hyperextension exercises of the thigh and trunk in an erect posture. Weakness of gluteal muscles causes decreased sacroiliac (SI) joint stability in patients with sacroiliac disorders. gluteus maximus muscle, due to its attachments to the sacrum, iliac bones, and sacrotuberous ligament, plays a significant role in the stability of the SI joint. The stabilizing forces applied to the SI joint, therefore, could be compromised with gluteal muscle weakness. In patients with gluteal weakness, shortening of the hamstring muscles, through their common attachments to the ischial tuberosity and sacrotuberous ligament, could compensate for gluteal muscle weakness and contribute to the SI joint stability.

A relationship between the gluteus maximus and the SI joint has been investigated in particular. Anatomical studies suggest that the gluteus maximus, with muscle fibers perpendicular to the joint surfaces, can help to stabilize the SI joint. Furthermore, it was discovered that activating the gluteus maximus increased compressive force across the SI joint. Individuals with SI joint dysfunction have abnormal gluteus maximus recruitment during weight-bearing exercises. As a result, it is hypothesized that gluteus maximus weakness can be linked to incorrect loading of the SI joint and be a cause of the impairments associated with SI joint dysfunction.

Hip extension exercise is the general clinical method for improving the weakened muscle strength of the hip extensors. These exercises are often used to strengthen the gluteus maximus and is also recommended for patients with pain in the lower back, pelvis, or hip. The gluteus maximus contributes to the postural alignments, core stability, and functional abilities that are important for normal gait. A weakness of the gluteus maximus can cause an abnormal gait cycle that can affect the gait mechanics at both hip and knee joints. In particular, gluteus maximus exercise is important for patients who have low back pain and lower extremity injuries. Patients with low back pain show reduced activity of the gluteus maximus. Early activation of the hamstring muscles and spinal erector, as well as delayed or decreased activation of the gluteal muscles, are considered indications of faulty muscle activation.

Studies have assessed methods for selective strengthening of the gluteus maximus. Prone hip extension (PHE) exercise is generally used to activate and strengthen the gluteus maximus selectively. Active prone hip extension with knee flexion is a common exercise employed to optimize gluteus maximus activation because this position causes active insufficiency of the hamstring. A previous study reported that PHE exercise is the most effective method for activating the gluteal muscles when subjects extend their hip with 30° abduction. Other studies have suggested that an abdominal drawing-in maneuver (ADIM) with prone hip extension is useful for the selective activation of the gluteus maximus from the erector spinae and hamstring.

A correction of the abnormal pattern is recommended to reduce the stress on the spine and hip joint. In a clinical setting, the ADIM is used during hip extension to prevent abnormal motion of the pelvis and lumbar., and the degree of knee extension affects the gluteus maximus activity. When the level of knee extension is increased, the activity of the gluteus maximus decreases, and the hamstring activity increases. Previous studies compared the muscle activities of the hamstring and gluteus maximus during prone hip extension with ADIM. The following were applied during active prone hip extension exercises: knee flexion, knee extension, hip external rotation with knee flexion, and hip external rotation with knee extension. In addition, eleven different exercises of the gluteus maximus used in therapeutic exercises were compared.

Although a wide variety of different exercises are advocated train and condition gluteus maximus and surrounding musculature, there are no specific guidelines for gluteus maximus strengthening with SI joint dysfunction using best evidence-based practice. This study aims to find out whether the weighted and elastic resistance training of gluteus maximus provides better results in subjects with SIJ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* pain in the SI region for at least 12 weeks (chronic) and had no previous physical therapy treatment
* SIJ dysfunction confirmed by tests described by McGrath et al.
* These tests included the SI compression, SI distraction, Squish, and Gaenslen.

Exclusion Criteria:

* Subjects with clinical and imaging evidence of any other spinal or pelvic co-morbidity potentially responsible for pain radiating through the sacroiliac region.
* True leg length discrepancy [measured from the anterior superior iliac spine (ASIS) to the medial malleolus.
* Back, pelvis, hip, or knee fracture history or surgery.
* Having a systemic pathology including inflammatory joint disease
* Having a musculoskeletal or neurological disease
* Having taken anti-inflammatory medication

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Gluteus maximus strength with a dynamometer | 5th week
  hand held dynamometer is placed over gluteus maximus in position of hip extension ad knee flexion and asked the patient to contract for three seconds against resistance nad record reading.
Oswestry disability index | 5th week
  This questionnaire consists of 10 sections describing the pain and its impact. Each section scores from 0 to 5, 0 being no pain and 5 being severe pain. The domains include pain intensity, personal care, lifting, sitting, walking, standing, sleeping, travel, social life, and change in the degree of pain.
Numeric Pain Rating Scale | 5th week
  this is scale for measuring pain. it is 11 point scale with 0 at no pain and 10 at max pain

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- King Abdullah Teaching Hospital, Mānsehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lingutla KK, Pollock R, Ahuja S. Sacroiliac joint fusion for low back pain: a systematic review and meta-analysis. Eur Spine J. 2016 Jun;25(6):1924-31. doi: 10.1007/s00586-016-4490-8. Epub 2016 Mar 8. PMID 26957096
- [Background] Selkowitz DM, Beneck GJ, Powers CM. Comparison of Electromyographic Activity of the Superior and Inferior Portions of the Gluteus Maximus Muscle During Common Therapeutic Exercises. J Orthop Sports Phys Ther. 2016 Sep;46(9):794-9. doi: 10.2519/jospt.2016.6493. Epub 2016 Aug 5. PMID 27494053
- [Background] Added MAN, de Freitas DG, Kasawara KT, Martin RL, Fukuda TY. STRENGTHENING THE GLUTEUS MAXIMUS IN SUBJECTS WITH SACROILIAC DYSFUNCTION. Int J Sports Phys Ther. 2018 Feb;13(1):114-120. PMID 29484248
- [Background] Bae C-H, Choe Y-W, Kim M-K. Effects of Different External Loads on the Activities of the Gluteus Maximus and Biceps Femoris during Prone Hip Extension in Healthy Young Men. Korean Society of Physical Medicine. 2020;15(2):1-9.